CLINICAL TRIAL: NCT02350010
Title: The Research of Etiology and Risk Factors Related to Prognosis of Intracerebral Hemorrhage in Beijing
Brief Title: Etiology and Prognostic Risk Factors of Intracerebral Hemorrhage in Beijing
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Neurosurgical Institute (Other)
Collaborators: Peking University Third Hospital (Other); Beijing Tiantan Hospital (Other); Beijing Shijitan Hospital, Capital Medical University (Other); KaiLuan General Hospital (Other); Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other); People's Hospital of Beijing Daxing District (Other); Beijing Aerospace General Hospital (Other); Beijing Haidian Hospital (Other); Beijing Fangshan District Liangxiang Hospital (Other); The 263 Hospital of PLA (Unknown); General Hospital of Beijing PLA Military Region (Other); Peking University Aerospace Center Hospital (Other); Beijing Renhe Hospital (Unknown); Beijing Pinggu District Hospital (Other); Beijing Shuyi Hospital (Other); Beijing Huairou Hospital (Other); Beijing Luhe Hospital (Other); Fu Xing Hospital, Capital Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: D141100000114003
Record Dates: First submitted 2015-01-07; First posted 2015-01-29 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Intracerebral Hemorrhage
Keywords: Etiology; Prognostic risk factors; Intracerebral Hemorrhage; non-invasive imaging; CT angiography
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Computed Tomography Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: CT Angiography — CTA Scan with the specified sequences below:
  120 kVp, 360 mAs, 0.5 second/rotation, 0.75 mm thick with a pitch of 0.65. Coronal and sagittal multiplanar reconstructed images with 10.0-mm-thick images spaced by 3 mm.
  Axial reformed images were 4 mm thick with 2-mm spacing. 90 mL of nonionic iodinated contrast (OPTIRAY 350) at 5 mL/s.

SUMMARY:
There were lack of data and analysis about medical management, etiology, and long-term outcome of Intracerebral Hemorrhage (ICH) in Beijing. In this study the investigators do acute CT angiography, a non-invasive imaging method to explore etiology and prognostic risk factors of ICH. Further the investigators will aim to develop and validate a risk score for predicting 1-year functional outcome after ICH.

DETAILED DESCRIPTION:
Intracerebral hemorrhage (ICH) accounts for 10 %-15 % of all strokes and is one of leading causes of stroke related mortality and morbidity worldwide. Despite advances in medical knowledge, treatment for ICH remains strictly supportive. ICH accounted for 26.7～51.5% of stroke in China, the proportion was higher than in Western countries. There were lack of data and analysis about medical management, etiology, and long-term outcome of ICH in Beijing.

In this study we do acute CT angiography (CTA), a non-invasive imaging method to explore etiology and prognostic risk factors of ICH. Further we will aim to develop and validate a risk score for predicting 1-year functional outcome after ICH. There are some studies of CTA to assess the cause of ICH and functional outcomes, but lack of multi-center, large sample studies to support and validate these findings, particularly fewer application of postcontrast CT. This would allow an early intervention base on different causes and Select treatment decisions according to risk score.

We are planning to:

When patients with ICH arrive in stroke department of the topic cooperation hospitals within 72 hours after symptom onset, they will be subject to CTA with the protocoled sequences.

Standard sequences: Pre- and postcontrast head imaging is acquired from the skull base to vertex with parameters: 120 kVp; 340 mA; 4x5 mm collimation; 1second/rotation; and a table speed of 15 mm/rotation. CTA was performed immediately after initial noncontrast CT(NCCT) performance using a bolus-tracking method by injecting 90 mL of nonionic iodinated contrast (OPTIRAY 350) at 5 mL/s. The protocol for the circle of Willis was 120 kVp, 360 mAs, 0.5 second/rotation, 0.75 mm thick with a pitch of 0.65. Postprocessing procedure including multiplanar reconstruction was performed by a CT technologist at the CT operator's discretion for assessment of contrast extravagation and etiologies of ICH such as vascular malformation, and venous sinus thrombosis. Coronal and sagittal multiplanar reconstructed images were created as 10.0-mm-thick images spaced by 3 mm. Axial reformed images were 4 mm thick with 2-mm spacing.

Clinical data of patients with ICH will be collected by 2 neurologists blinded to the radiological data during patients' hospitalization and at the 3-month, 6-month, and 1-year follow-up. The collected demographic and clinical variables included gender, age, body mass index, alcohol and tobacco use, history of hypertension, diabetes, hyperlipidemia, stroke, coronary heart disease, and medications (antihypertensive, antiplatelet, and anticoagulation agents). The systolic and diastolic blood pressure of patients will be recorded. Stroke severity on admission will be evaluated by Glasgow Coma Scale and National Institutes of Health Stroke Scale. Laboratory tests on admission included white blood cell count, hemoglobin, platelet count, serum glucose, serum creatinine, fibrinogen, activated partial thromboplastin time, and prothrombin time as expressed by the international normalized ratio. Length of hospital stay was recorded. The patients' clinical outcome will be assessed by modified Rankin Scale on discharge and 30-day, 3-month, 6-month, and 1-year.

To sum up the purpose of this present study is to explore etiology and prognostic risk factors of ICH by acute CTA and develop and validate a risk score for predicting 1-year functional outcome after ICH.

ELIGIBILITY:
Inclusion Criteria:

* CT demonstrated ICH
* Age above 18
* within 72 hours of symptom onset
* Informed consent from patient or proxy

Exclusion Criteria:

allergy to contrast medium incompletion of a standard CT protocol including noncontrast CT (NCCT) and CTA Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted with CT-demonstrated Intracerebral Hemorrhage (ICH) within 72 hours after symptom onset.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
one-year functional outcome and mortality of Intracerebral hemorrhage. | one year
  Good functional outcome was defined as modified Rankin Scale score (mRS) ≤2.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Zhi Wang, professor, Study Chair — Beijing Neurosurgical Institute
Locations (1):
- Beijing Neurosurgical Institute, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Hemphill JC 3rd, Bonovich DC, Besmertis L, Manley GT, Johnston SC. The ICH score: a simple, reliable grading scale for intracerebral hemorrhage. Stroke. 2001 Apr;32(4):891-7. doi: 10.1161/01.str.32.4.891. PMID 11283388
- [Background] Hemphill JC 3rd, Farrant M, Neill TA Jr. Prospective validation of the ICH Score for 12-month functional outcome. Neurology. 2009 Oct 6;73(14):1088-94. doi: 10.1212/WNL.0b013e3181b8b332. Epub 2009 Sep 2. PMID 19726752
- [Background] Feigin VL, Lawes CM, Bennett DA, Barker-Collo SL, Parag V. Worldwide stroke incidence and early case fatality reported in 56 population-based studies: a systematic review. Lancet Neurol. 2009 Apr;8(4):355-69. doi: 10.1016/S1474-4422(09)70025-0. Epub 2009 Feb 21. PMID 19233729
- [Background] van Asch CJ, Luitse MJ, Rinkel GJ, van der Tweel I, Algra A, Klijn CJ. Incidence, case fatality, and functional outcome of intracerebral haemorrhage over time, according to age, sex, and ethnic origin: a systematic review and meta-analysis. Lancet Neurol. 2010 Feb;9(2):167-76. doi: 10.1016/S1474-4422(09)70340-0. Epub 2010 Jan 5. PMID 20056489
- [Background] Zhang LF, Yang J, Hong Z, Yuan GG, Zhou BF, Zhao LC, Huang YN, Chen J, Wu YF; Collaborative Group of China Multicenter Study of Cardiovascular Epidemiology. Proportion of different subtypes of stroke in China. Stroke. 2003 Sep;34(9):2091-6. doi: 10.1161/01.STR.0000087149.42294.8C. Epub 2003 Aug 7. PMID 12907817
- [Background] Jiang B, Wang WZ, Chen H, Hong Z, Yang QD, Wu SP, Du XL, Bao QJ. Incidence and trends of stroke and its subtypes in China: results from three large cities. Stroke. 2006 Jan;37(1):63-8. doi: 10.1161/01.STR.0000194955.34820.78. Epub 2005 Nov 23. PMID 16306469
- [Background] Morgenstern LB, Hemphill JC 3rd, Anderson C, Becker K, Broderick JP, Connolly ES Jr, Greenberg SM, Huang JN, MacDonald RL, Messe SR, Mitchell PH, Selim M, Tamargo RJ; American Heart Association Stroke Council and Council on Cardiovascular Nursing. Guidelines for the management of spontaneous intracerebral hemorrhage: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2010 Sep;41(9):2108-29. doi: 10.1161/STR.0b013e3181ec611b. Epub 2010 Jul 22. PMID 20651276